CLINICAL TRIAL: NCT06632782
Title: A Pilot Study to Assess the Impact of Breath Awareness Using Pyramid on Symptoms of Anxiety and Depression in People with T2DM
Acronym: BAPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dasman Diabetes Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RA HM 2023-001
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Depression, Anxiety
Keywords: depression
MeSH Terms: conditions — Depression; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomized to the intervention and control group.
Who Masked: Investigator
Masking Description: Masking of participants is not possible in such alternative intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intervention (Experimental): Breath Awareness using pyramid in people with T2DM and symptoms of depression and anxiety
  Interventions: Behavioral: Breath Awareness using pyramid
- control (No Intervention): Control group or the wait list group will continue usual treatment recommended by the physician.

INTERVENTIONS:
Behavioral: Breath Awareness using pyramid — Participants are provided 1-2 hr training for 6 weeks on bringing breath awareness to the present moment using a pyramid
  Other Names: mindfulness
  Arms: intervention

SUMMARY:
Diabetes mellitus is rampant in the Middle East. It is a psychologically and behaviorally demanding disease; psychosocial factors are relevant to nearly all aspects of its management. Moreover, depression and diabetes are bidirectionally connected. Those with depression are at risk of developing diabetes and those with comorbid diabetes are at risk of developing depressive symptoms. Research findings have demonstrated that depression and anxiety are more common in patients with diabetes than in the general population, atleast 15 % have clinical depression. In addition, the recent COVID- 19 pandemic has fueled the burden by increasing fear, anxiety, and depression among people with T2DM due to susceptibility to long-term complications. In Kuwait, a recent survey found the prevalence of depression to be 29% and diabetes distress to be 14%. Thus, there is a dire need to address this challenging problem. In the recent past, mindfulness-based intervention such as Mindfulness-based stress reduction (MBSR), Mindfulness-based cognitive therapy (MBCT,) and yoga have emerged as unique tools for reducing a wide range of psychological disorders. These tools positively impact hormone regulation and have a beneficial effect on cognitive function and increased parasympathetic activity. The positive impact of mindfulness is assumed to be amplified if a pyramid structure with geometry similar to the pyramid of Giza is used for practice. Not much human research has been performed to demonstrate that pyramid energy along with mindfulness can be a tool to combat psychological disorders. However, few studies on animal models provided evidence of the potential beneficial effect of pyramid structure in reducing stress. Previous pilot study conducted using only yoga as an intervention indicated significant improvement in anxiety, depression, and quality of life in people with T2DM. However, there was no change in participants' glycemic control. In this pilot study, investigator will assess whether pyramid breath awareness can alleviate symptoms of depression and anxiety in people with T2DM.

DETAILED DESCRIPTION:
Hypothesis of the study is whether the combination of breath awareness and pyramid energy will

* Amplify the positive impact on mental health in people with T2DM
* Impact the glycaemic control in people with T2DM Methodology: Experimental Design

This is a randomized controlled trial study to assess the effect of pyramid breath awareness on people with T2DM and symptoms of depression. Eligible participants will be randomly assigned to either the interventional group or the waitlisted group (control group) in a ratio of 1:1. The participants in the intervention group will be provided with a training session on breath awareness using a pyramid head cap. Participants in the waitlisted group (control group) will be following the usual care recommended by the physician. However, breath awareness training will be given to the waitlist group after the study.Hospital Anxiety and Depression Scale (HADS), the Patient Health Questionnaire (PHQ-9), the Perceived Stress Scale, Diabetes Quality of Life (DQoL), the Pittsburgh Sleep Quality Index (PSQI), and the Mindful Attention Awareness Scale (MAAS) at baseline, 6th week and 12th week. 12 ml of blood will be drawn from the participants of both groups by a trained phlebotomist. Participants in the intervention group will be provided with breath awareness training by a certified breath awareness trainer. Participants will be instructed to be aware of their breath by placing the pyramid cap on their head. Apart from breath awareness technique, group discussion on healthy, mindful living, and wisdom sharing will be carried out by the trainer. A total of 1 to 2 hours of daily sessions will be provided to the participants until 6 weeks at DDI or online as preferred by them, followed up until 12 weeks later. The compliance rate of participants will be monitored using an attendance log. Participants glycaemic control (HbA1C), cortisol, lipid profile, TSH, complete clinical report, and other inflammatory biomarkers will be measured at three intervals, baseline, 6th week, and 12th week.

Statistical method: Sample Size Calculation: Based on the previous studies and a prevalence of 29 % depression in the state of Kuwait, sample size of 76 is considered for the pilot study. 25% more will be recruited to account for dropouts and defaulter. Data management: Data will be collected by a trained research team and will be entered into the REDCAP with proper scrutiny and quality checks.The data will be kept confidential, and the team will ensure good documentation and assure to comply with good clinical practices. The team members are GCP trained and will undergo online training provided by CITI.

ELIGIBILITY:
Inclusion Criteria: • More than 1 year of T2DM diagnosis

* T2DM with HbA1c greater than 5.7 and less than 9.5%
* T2DM patients, age greater than 30 years and on oral hypoglycaemic agents or on insulin
* No cardiac problems
* Score 8.0 and above as per the anxiety and depression questionnaires.
* Able to be aware of breath and provide written informed consent.

Exclusion Criteria:

* T1DM patients
* On antidepressant drugs
* Bipolar disorders
* Any acute coronary events in the past 6 months
* Any acute renal diseases including transplant or dialysis.
* Artificial pacemaker
* Any breath awareness or yoga course within 6 months.
* Pregnancy

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Hospital Anxiety and depression score(HADS) | 6 weeks
  HADS is assessed at baseline and at 6th Week to assess anxiety and depression. A lower score indicates a better outcome(less than 8).
Change in Patient Health Questionnaire PHQ-9 score | 6 weeks
  PHQ-9 score is assessed at baseline and at 6th week to assess depression, lower score indicates a better outcome(less than 4)
Change in Pitssburgh Sleep Quality Index PSQI score | 6 weeks
  PSQI score is assessed at baseline and in 6th week to assess the sleep quality, less than 5 indicate better outcome
Change inMindful Attention Awareness Scale (MAAS) | 6 weeks
  MAAS score is measured at baseline and in 6th week to assess the mindfulness. Higher score indicate better outcome

SECONDARY OUTCOMES:
Change in Diabetes Quality of Life (Diabetes 39) | 6 weeks
  DQoL score is measured at baseline and in 6th week to assess the quality of life.
Change in HbA1C | 6 weeks
  HbA1c is measured at baseline and in 6th week to assess the glycemic control
Change in cortisol levels | 6 weeks
  Serum cortisol level is measured at baseline and in 6th week to assess the stress indicator

CONTACTS AND LOCATIONS:
Overall Officials: Rashmi Shiju, Principal Investigator — Dasman Diabetes Institute
Locations (1):
- Dasman Diabetes Institute, Kuwait City, Kuwait, Kuwait